CLINICAL TRIAL: NCT00795158
Title: An Open-Label Study of the Effects of Desloratadine Treatment on the Quality of Life of Patients With Chronic Urticaria
Brief Title: How Desloratadine (Clarinex, Aerius) Affects Quality of Life in Patients With Chronic Idiopathic Urticaria (Have Had Hives for 6 Weeks or Longer)(Study P02988)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02988
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Urticaria
MeSH Terms: conditions — Urticaria | interventions — desloratadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: desloratadine

INTERVENTIONS:
Drug: desloratadine — desloratadine 5 mg tablets; one tablet orally once a day for 28 days
  Other Names: Clarinex; Aerius; SCH 34117; descarboethoxyloratadine

SUMMARY:
The purpose of this study was to determine the effect of desloratadine treatment on quality of life, daytime functioning, quality of sleep, symptoms, and disease severity in patients who had hives for 6 weeks or longer. Patients took desloratadine for 1 month. Once a week, patients filled out a questionnaire to tell how their hives affected their lives. This questionnaire is called the Dermatology Life Quality Index or DLQI. They also filled out a diary every day to tell how much itching they had, how many hives they had, and how their hives had affected their sleep or daily activities. The patients and doctors rated the patients' overall condition and how much relief patients got from treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must demonstrate their willingness to participate into the study and comply with its procedures by signing a written informed consent.
* Subjects must be >=18 years of age, of either sex and any race.
* Women of childbearing potential (includes women who are less than 1 year postmenopausal) must be using an acceptable method of birth control since at least one month prior to visit 1 (e.g., hormonal contraceptive, medically prescribed IUD, condom in combination with spermicide) or be surgically sterilized (e.g., hysterectomy or tubal ligation). Women of childbearing potential should be counseled in the appropriate use of birth control while in this study.
* Subjects must be in general good health as confirmed by medical history and, physical examination; i.e., they must be free of any clinically significant disease (other than chronic urticaria [CU]) that would interfere with study evaluations.
* Subjects must understand and be able to adhere to the dosing and visit schedules, and agree to complete the questionnaires and to record accurately and consistently in a daily diary symptom severity scores, medication times, concomitant medications, and adverse events.
* Subjects must have a history of CU defined as at least 6 weeks of pruritus and hives with hives lasting less than 24 hours and occurring at least 2 days per week.
* Subjects must be experiencing a current CU flare with hives present at least 2 days in the week prior to the consent visit/visit 1.
* Subjects must have a pruritus score >=2 and a hive score >=1 at consent visit/Visit 1 or during the 12 hours before the consent visit/Visit 1
* Subjects must score the Overall Condition of CU >=2 at both consent visit/Visit 1 and Visit 2 (Baseline).
* Subjects must have a total pruritus score of >=11 for the sum of morning (AM) and evening (PM) (reflective) diary scores for the 3 days prior to Visit 2 (Baseline) plus the morning score on the day of Visit 2
* Women of childbearing potential must have a negative urine pregnancy test at Visit 2 (Baseline).

Exclusion Criteria:

* Women who are pregnant or nursing.
* Subjects who have not observed the designated washout periods for any of the prohibited medications
* Subjects with asthma
* Subjects with drug or food allergies that manifest as skin reactions during 1 year prior to consent visit / visit 1
* Subjects with atopic dermatitis
* Subjects with urticaria that is primarily due to physical urticaria or other known etiology (on the basis of clinical history and physical examination).
* Subjects with CU unresponsive to antihistamines.
* Subjects under regular treatment with NSAIDs.
* Subjects who have been hospitalized because of worsening in their CU within 3 months prior to Visit 1 (Screening).
* Subjects with a history of hypersensitivity to Desloratadine or any of its excipients.
* Subjects previously enrolled into this study (i.e. who have been assigned to treatment).
* Subjects who are staff personnel directly involved with the administration of this study.
* Subjects who have any clinically significant metabolic, cardiovascular, immunologic, neurologic, hematologic, neoplastic, gastrointestinal, cerebrovascular, or respiratory disease, or any other disorder which, in the judgment of the Investigator, may interfere with the study evaluations or affect subject safety.
* Subjects with a history of psychosis, antagonistic personality, poor motivation, hypochondriasis, or any other emotional or intellectual problems that are likely to limit the validity of consent to participate in the study.
* Subjects with a history of noncompliance with medications or treatment protocols.
* Subject treated with any investigational drug in the last 30 days prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2002-11; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to day 28 in Dermatology Life Quality Index (DLQI) score | Baseline and treatment day 28

SECONDARY OUTCOMES:
Change from Baseline in the DLQI score on treatment days 7, 14, 21 | Baseline and treatment days 7, 14, 21
Change from Baseline in pruritus, the number of hives, sleep quality, and daily activity impairment on treatment days 7, 14, 21, and 28 | Baseline and treatment days 7, 14, 21, and 28
Change from Baseline in the Overall Condition of chronic urticaria on treatment days 14 and 28 | Baseline and treatment days 14 and 28
Percent of subjects who rate their response to therapy as either Complete, Marked, or Moderate Relief on treatment days 14 and 28 | Treatment days 14 and 28
Evaluation of tolerability and safety by clinical laboratory tests | Baseline and treatment day 28
Evaluation of tolerability and safety by adverse events | Screening, Baseline, and treatment days 14 and 28

REFERENCES:
- [Result] Seidenari S, Cirillo A, Amoroso S, Flori ML, Amerio P, Ricciuti E, Vena GA, Berardesca E, Le Grazie C and the Italian Study Group on Desloratadine (DL) in Chronic Urticaria. Desloratadine 5 milligrams once daily improves quality of life in chronic idiopathic urticaria. G Ital Dermatol Venereol. 2006;141(3):207-214